CLINICAL TRIAL: NCT05764564
Title: External Body Pressure and the Impact on Exercise in Heart Failure With Preserved Ejection
Brief Title: External Body Pressure in Heart Failure With Preserved Ejection Fraction
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00112081
Record Dates: First submitted 2023-02-25; First posted 2023-03-10 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-02

CONDITIONS: Heart Failure, Diastolic
MeSH Terms: conditions — Heart Failure, Diastolic | interventions — Gene Expression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Experimental: Patients with heart failure (Aim 1) (Experimental)
  Interventions: Diagnostic Test: Positive or negative pressure
- Control: Healthy Volunteers (Aim 1) (Active Comparator)
  Interventions: Diagnostic Test: Positive or negative pressure
- Experimental: Patients with heart failure (Aim 2) (Experimental)
  Interventions: Diagnostic Test: Positive or negative pressure

INTERVENTIONS:
Diagnostic Test: Positive or negative pressure — Positive or negative pressure is applied via a closed chamber.

SUMMARY:
The primary objective of the study is to test the impact of positive and negative body pressure on exercise capacity, symptoms, blood volume distribution and central cardiac hemodynamics in patients with heart failure and preserved ejection fraction. Aim 1 will study healthy volunteers and heart failure patients non invasively while Aim 2 will study heart failure patients invasively (intracardiac pressures).

ELIGIBILITY:
* Heart Failure Study Population
* Inclusion Criteria (Aim 1 and 2):

  * Age greater than or equal to 30 yrs
  * Established diagnosis of HFpEF with left ventricular ejection fraction greater than or equal to 50%
  * NYHA II-III symptoms
  * Stable HF drug regimen for the preceding 1 month
  * Wedge pressure greater than or equal to 15 mmHg at rest or greater than or equal to 25 mmHg with peak exercise
  * (For Aim 2 only) Scheduled for an elective right heart catheterization at Duke University Hospital.
* Exclusion Criteria (Aim 1 and 2):

  * HF hospitalization for type I myocardial infarction within 3 months
  * Infiltrative (ie amyloid) or hypertrophic cardiomyopathy
  * Uncontrolled atrial or ventricular arrhythmia
  * Chronic oxygen use
  * History of vasovagal syncope
  * Considered inappropriate to participate by PI or Sub-I
  * Healthy Volunteers (Controls)
* Inclusion Criteria (Aim 1):

  * Age greater than or equal to 30 yrs
  * Able to speak English
  * Ambulatory [assistive devices ok]
  * Able to provide informed consent
* Exclusion Criteria (Aim 1):

  * Acute myocardial infarction (3-5 days)
  * Unstable angina
  * Uncontrolled arrhythmia causing symptoms or haemodynamic compromise
  * Syncope
  * Active endocarditis
  * Acute myocarditis or pericarditis
  * Symptomatic severe aortic aneurysm
  * Uncontrolled asthma
  * Arterial desaturation at rest on room air <85%
  * Untreated left main stem coronary stenosis
  * Asymptomatic severe aortic stenosis
  * Severe untreated arterial hypertension at rest (>200 mm Hg systolic, >120 mm Hg diastolic)
  * Tachyarrhythmias or bradyarrhythmias
  * Hypertrophic cardiomyopathy
  * Significant pulmonary hypertension
  * Thrombosis of the lower extremity until treated for a minimum of 2 weeks
  * Within 2 weeks of acute symptomatic pulmonary embolus
  * Abdominal aortic aneurysm >8.0 cm
  * Electrolyte abnormalities
  * Pregnancy
  * Inmate of correctional facility (i.e. prisoner)
  * Diagnosed history of dementia
  * Inability to ambulate independently
  * Considered inappropriate to participate by Principal Investigator

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2023-04-21 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
change in exercise cardiac output | Day 1
  Change in cardiac output from rest to 0 Watts exercise

SECONDARY OUTCOMES:
change in exercise cardiac output | Day 1
  Change in cardiac output from rest to 20 Watts exercise
change in heart rate | Day 1
  Change in heart rate from rest to 0 Watts exercise
change in heart rate | Day 1
  Change in heart rate from rest to 20 Watts exercise
change in respiratory rate | Day 1
  Change in heart rate from rest to 20 Watts exercise
change in O2 consumption | Day 1
  Change in O2 consumption from rest to 0 Watts exercise
change in O2 consumption | Day 1
  Change in O2 consumption from rest to 20 Watts exercise
Change in wedge pressure | Day 1
  Change in wedge pressure from rest to 0 Watts exercise
Change in wedge pressure | Day 1
  Change in wedge pressure from rest to 20 Watts exercise

OTHER OUTCOMES:
Symptom burden | Day 1
  from rest to peak exertion we will assess symptom burden with dyspnea scales

CONTACTS AND LOCATIONS:
Overall Officials: Hemming, Study Chair — Duke
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No